CLINICAL TRIAL: NCT03695666
Title: A Completed-cycle Local Audit of Patient Load in the SHO-led ENT Casualty Clinic
Status: Completed | Type: Observational
Sponsor: National Health Service, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Sadik Quoraishi, PI, National Health Service, United Kingdom
Other Study IDs: w106k6eMBibC
Record Dates: First submitted 2018-10-01; First posted 2018-10-04 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: ENT Disease
MeSH Terms: conditions — Otorhinolaryngologic Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cycle 1: Counted number of patients booked into clinic. No individual patient data collected.
- Cycle 2: Counted number of patients booked into clinic. No individual patient data collected.
  Interventions: Other: Clerical policy

INTERVENTIONS:
Other: Clerical policy — Clerical policy introduction
  Groups: Cycle 2

SUMMARY:
ENT UK guidelines recommend booking no more than 6 patients during each 4-hour clinic session. Retrospectively, the investigators counted patients booked for each clinic on ourbooking system. The second cycle showed improved compliance with guidelines.

DETAILED DESCRIPTION:
Background The investigators' centre runs a regular ENT casualty clinic, run by an SHO, for rapid assessment and treatment of simple, acute ENT cases. ENT UK guidelines from 2017 recommend that no more than 6 patients be booked for an SHO to see during a 4-hour clinic session. This study aims to assess whether this centre meets those guidelines.

Method Data was retrospectively collected from MedWay, the centre's networked booking system. The number of patients booked for each ENT casualty clinic was counted over a period of two months. This was repeated two months after intervention to close the loop.

Result In the first cycle, 2 out of 22 clinics (9%) were found to be compliant with guidelines. Our intervention was to inform clinic booking staff of the guidelines. In the second cycle, 20 of 24 clinics were compliant (83%).

Discussion Anecdotally, prior to intervention, SHOs would often struggle to keep up with the casualty clinic caseload, and clinics would overrun. Clinic booking staff were not previously aware of ENT UK guidelines, and the number of clinic slots was set arbitrarily. This was easily and effectively resolved by educating staff. It can be learned that de facto management practice is not always based on guidelines or evidence; and highlights the importance of auditing all aspects of how organisations are run. Further quality improvement studies should focus on what happens to patients who can no longer be fit into existing casualty clinics.

ELIGIBILITY:
Inclusion Criteria:

* All ENT casualty clinics with patients booked within the study time period

Exclusion Criteria:

* All clinics that were not staffed by an SHO

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients booked into SHO-led ENT casualty clinics
Sampling Method: Non-Probability Sample
Enrollment: 333 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-03-14 (Actual); Study Completion 2018-03-14 (Actual)

PRIMARY OUTCOMES:
Retrospectively counted patients booked | 2 months
  Retrospectively counted patients booked

CONTACTS AND LOCATIONS:
Overall Officials: Sadik Quoraishi, Principal Investigator — National Health Service, United Kingdom
Locations (1):
- Royal Stoke University Hospital, Stoke-on-Trent, United Kingdom

IPD SHARING:
Plan to Share IPD: No